CLINICAL TRIAL: NCT02676362
Title: Methodological Evaluation of Gingival Crevicular Fluid Volume and Elastase Levels: Sequential Sampling, Length of Sampling Time And Two Different Sampling Methods
Brief Title: Methodological Evaluation of Gingival Crevicular Fluid Volume and Elastase Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nilgün Özlem Alptekin, Prof., DDS, PhD, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 08/05
Record Dates: First submitted 2016-02-01; First posted 2016-02-08 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- the first day (Experimental): Gingival crevicular fluid collection with filter paper the length of sampling time in seconds: 5., 10., 30.
  Interventions: Other: Gingival crevicular fluid collection with filter paper
- the 2nd day (Experimental): Gingival crevicular fluid collection with filter paper the length of sampling time in seconds: 10., 30., 5.
  Interventions: Other: Gingival crevicular fluid collection with filter paper
- the 3rd day (Experimental): Gingival crevicular fluid collection with filter paper the length of sampling time in second: 30., 5., 10.
  Interventions: Other: Gingival crevicular fluid collection with filter paper

INTERVENTIONS:
Other: Gingival crevicular fluid collection with filter paper — Gingival Crevicular Fluid Dynamics

SUMMARY:
The mechanisms underlying the formation and composition of gingival crevicular fluid (GCF) and its flow into and from periodontal pockets are not understood very well. The aim of this study was to evaluate the length of sampling time and sequential sampling of GCF neutrophil elastase (NE) enzyme activity by using intracrevicular and orifice methods.

DETAILED DESCRIPTION:
Twenty adults (mean age of 41.8 years. ranged 31-60 years. 18 males. 2 females) with chronic periodontitis were enrolled and all completed the 3-day study. Three-hundred-sixty samples of GCF were harvested from the interproximal sites of each of the two maxillary non-molar teeth according to the orifice method. Each site was sampled three times with 1-min intervals between repeat samples. By using intracrevicular method, the other 360 samples of GCF were collected on the same sites following 10-minutes interval. In first day, 2nd day and 3rd day the length of sampling time in seconds and order were 5. 10. 30; 10. 30. 5 and 30. 5. 10. respectively. GCF elastase activity was determined by hydrolysis of neutrophil specific substrate N-methoxysuccinyl-Ala-Ala-Pro-Val-p-nitroanilide and was expressed as concentration (microU/microl) and total enzyme activity (microU).

ELIGIBILITY:
Inclusion Criteria:

* no history of systemic disease;
* no history of antibiotics and/or anti-inflammatory drugs within the past 6 months;
* no received any oral hygiene prophylaxis and scaling and root planing within the past 6 months;
* at least 2 interproximal sites exhibiting higher than 5 mm probing depth, radiographic bone loss and gingival index of 2 (with preference of two maxillary non-molar teeth)

Exclusion Criteria:

* with metabolic diseases
* pregnancy, lactation etc.

Ages: 31 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The length of sampling time of GCF Elastase Levels | 3 days

SECONDARY OUTCOMES:
The length of sampling time of GCF Volume | 3 days
The length of sequential sampling of GCF Volume | 3 days
The length of sequential sampling of GCF Elastase Levels | 3 days

IPD SHARING:
Plan to Share IPD: Yes